CLINICAL TRIAL: NCT05988762
Title: The Impact of Supramaximal Walkouts on Subsequent Back Squat Performance
Brief Title: Supramaximal Walkouts and Back Squat Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Michael J. Ormsbee, Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: STUDY00004217
Record Dates: First submitted 2023-07-28; First posted 2023-08-14 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Muscular Strength; Exercise Performance; Squat

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not be told whether they are performing the supramaximal or submaximal walkout. Black trash bags will be used to cover the weights during the walkout set so that the participant cannot see which condition they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supramaximal Walkout (Experimental): Walkout set performed at 110% 1RM
  Interventions: Other: Supramaximal Walkout
- Control (Submaximal Walkout) (Experimental): Walkout set performed at 30% 1RM
  Interventions: Other: Submaximal Walkout

INTERVENTIONS:
Other: Supramaximal Walkout — Walkout set performed at 110% 1RM. Participant will unrack the weight, step back and brace as if to perform a back squat, hold for 10 seconds, then re-rack the weight without performing the squat.
  Arms: Supramaximal Walkout
Other: Submaximal Walkout — Walkout set performed at 30% 1RM. Participant will unrack the weight, step back and brace as if to perform a back squat, hold for 10 seconds, then re-rack the weight without performing the squat.
  Arms: Control (Submaximal Walkout)

SUMMARY:
The goal of this randomized, counterbalanced, crossover study is to determine the effectiveness of performing a supramaximal walkout on enhancing subsequent back squat performance in trained lifters. The main question we aim to answer is whether bar velocity, power output, perceived exertion, and muscle activation are altered when performing the back squat exercise after a supramaximal walkout. On the first visit, participants will be informed of the study protocols before providing oral and written informed consent. Afterwards, participants will complete maximum voluntary isometric contraction (MVIC) testing for the quadriceps and gluteus maximus muscle groups to generate a normalization for the electromyography (EMG) measurements. During the second visit, participants will perform a 1RM back squat. The third and fourth visits will be the experimental visits, where they will perform either a supramaximal (110% 1RM) or submaximal (control; 30% 1RM) walkout. A set of 1 back squat at 92.5% 1RM will be performed prior to the walkout to serve as a baseline, then 3 sets of 1 at 92.5% 1RM will be performed afterwards.

DETAILED DESCRIPTION:
Initial Visit Participants will be asked to arrive at the Institute of Sports Sciences & Medicine (ISSM) following a 3 h fasting period having abstained from alcohol for the previous 24 h and heavy lower body exercise for the previous 48 h. Participants will then be informed of the study protocols and procedures before providing oral and written informed consent. Following the signing of the informed consent document, participants will complete the PAR-Q+ to determine readiness for physical activity and an additional training history form to assess their previous experience with exercise and resistance training. After completion of these documents, participants' blood pressure will be assessed via an automatic blood pressure monitor (Omron, Kyoto, Japan). Next, height will be assessed to the nearest cm using a wall-mounted scale (Seca, Hamburg, Germany). Participants will then be weighed to the nearest 0.1 kg via an automated scale (Detecto® 750, Webb City, MO). Body composition will then be assessed via BodPod (Cosmed, Chicago, IL).

Following these baseline measurements, surface electromyography (EMG) will be used to assess muscle activation. EMG electrodes (Noraxon, Arizona, USA) will be placed on the gluteus maximus and vastus lateralis muscle groups of the participants' dominant side to measure electrical potentials generated. Once the electrodes are in place, participants will complete a 5-min warmup on a cycle ergometer at a self-selected easy to moderate intensity before beginning maximum voluntary contraction (MVC) testing on an isokinetic dynamometer (Biodex Multi-Joint System-PRO, Biodex Medical Systems, Inc., Shirley, NY, USA). Isometric knee extension MVC torque will be measured with the knee joint flexed. The participant will test the isometric measurement three times at submaximal levels, followed by three maximal isometric contractions. Each contraction will last for 6 s and will be followed by 30 s rest. EMG amplitudes generated during this contraction will be used for EMG normalization. Following the testing on the dynamometer, participants will complete EMG normalization testing for the gluteus maximus. To determine this, participants will lie prone on a bench with their dominant knee flexed to 90°. Manual resistance will be applied to the distal thigh as the participant is instructed to extend their hip. Similar to the dynamometer testing, the participant will complete three submaximal repetitions followed by three maximal repetitions.

Preliminary Visit For the preliminary visit, participants will arrive to the ISSM having abstained from alcohol for the previous 24 h and heavy lower body exercise for the previous 72 h. Upon arrival, EMG electrodes will be applied to the same muscle groups as the initial visit. Participants will then complete a standardized warm up consisting of 5 min on the cycle ergometer at a self-selected easy to moderate pace, followed by a battery of dynamic movements (air squats, lunges, etc.) used to prepare the participant for the back squat exercise. Following this warm-up, participants will begin the 1RM back squat testing using a modified National Strength and Conditioning Association (NSCA) protocol. A linear position transducer system (Tendo Unit, Tendo Sports Machines, London, UK) will be attached to the barbell to evaluate bar velocity during the back squat movement. Following completion of the 1RM protocol, participants will perform a 5 min active recovery (cycle ergometer).

Experimental Visits For the experimental visits, participants will arrive to the ISSM a minimum of 72 h following the previous visit and having abstained from alcohol for the previous 24 h and heavy lower body exercise for the previous 72 h. Prior to testing, the EMG electrodes will be placed on the specific muscle groups and the linear position transducer will be attached to the barbell. The participants will begin by completing the same standardized warm up from the previous visit. After the standardized warm-up, participants will begin a specific warm-up with the back squat. The participant will first complete 8 repetitions at 30% of their target load (92.5% 1RM). After a 3 min rest, the participant will complete 5 repetitions @ 50% of their target load. After another 3 min rest, the participant will complete 3 repetitions at 70% of target load followed by another 3 min rest and the final warm-up set of 1 repetition @ 85% of target load. After a 5 min rest, the participants will then complete one repetition at 92.5% 1RM. Participants will be instructed to perform this set with maximum effort. Following a 5 min rest, the participants will then perform either the supramaximal or submaximal (control) walkout. Both walkouts will consist of the participant un-racking the bar and stepping back to get set up into their starting squat position. Instead of performing the squat, the participant will remain standing in place for 10 s before returning the bar to the rack. The supramaximal walkout will be performed at 110% 1RM while the control walkout will be performed at 30% 1RM. Before this walkout set, the weight on the bar will be covered with a black trash bag to blind the participant as to which trial they are in. This will negate any anticipatory effects leading up to the walkout. Then, immediately before the participant lifts the bar off the rack, the researchers will indicate whether the weight is light or heavy to avoid issues when un-racking the bar. After the walkout, the participant will rest for 5 min, followed by 3 sets of 1 repetition at 92.5% 1RM with 5 min rest between each set. Participants will be instructed to perform these sets at maximum velocity. Following the final set, participants will perform a 5 min active recovery (cycle ergometer).

Standardization of Diet and Training Prior to each experimental trial, participants will be asked to maintain consistent nutritional (dietary and supplementation) habits for the day preceding the experimental trial and the day of the experimental trial. Additionally, participants will be asked to avoid any lower body resistance exercise for the 72 h leading up to the experimental trial. To ensure compliance, participants will be asked to complete a 48-h dietary intake form (attached) and a 72-h exercise log (attached) for the days preceding the experimental trial. Finally, participants will be asked to abstain from any alcohol for 24 h prior to the experimental trial.

Bar Velocity, Muscle Activation, and RPE Peak and mean bar velocity (m/s) and power output (W) will be assessed via a linear position transducer system (Tendo Sport Machines, Trencin, Slovakia). The transducer system will be attached to the barbell prior to the onset of the specific warm-up. The measurement will be made independently for each set and automatically converted into values of peak power output and peak velocity.

Surface electromyography (EMG) will be used to assess muscle activation during each set of back squats. EMG electrodes (Noraxon, Arizona, USA) will be placed on the vastus lateralis and gluteus maximus of the participants' dominant side after the skin is shaved, abraded, and cleaned. The electrodes will be positioned longitudinally on the belly of each muscle. Data will be collected telemetrically at 1000 Hz and subjected to full-wave rectification. Baseline maximum EMG will be assessed during the maximal isometric torque assessment of the initial visit. EMG data collected during the back squat sessions will be normalized to the baseline EMG and presented as a percentage.

Rating of perceived exertion (RPE) will be assessed using a modified Borg RPE scale (attached). The participants will be familiarized with the scale prior to beginning the 1RM protocol.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male
* Age: 18-45 yr
* 1RM Back Squat ≥ 1.5x Body Weight

Exclusion Criteria:

* Musculoskeletal injuries limiting exercise capacity
* Cardiometabolic diseases limiting exercise capacity
* Hasn't performed squats in the past six months
* History of Rhabdomyolysis
* Use of anabolic steroids in the past year

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Back Squat Velocity | Baseline (5 minutes before walkout) and immediately after the walkout (3 sets with 5 minutes rest in between each set)
  Peak and average concentric bar velocity (m/s)
Back Squat Power Output | Baseline (5 minutes before walkout) and immediately after the walkout (3 sets with 5 minutes rest in between each set)
  Peak and average concentric power output (W)
Perceived Effort of Back Squat | Baseline (5 minutes before walkout) and immediately after the walkout (3 sets with 5 minutes rest in between each set)
  Rating of perceived exertion (RPE; 1-10)
Muscle Activation during Back Squat | Baseline (5 minutes before walkout) and immediately after the walkout (3 sets with 5 minutes rest in between each set)
  Electromyography (EMG) Amplitude

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ormsbee, PhD, Study Chair — Florida State University
Locations (1):
- Institute of Sports Sciences & Medicine, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Griest TD, McCarthy CM, Renteria LI, Paterson KGP, Eurich DF, Laskin GR, Ormsbee MJ. Supramaximal Walkouts Protect Against Performance Decrements Experienced in Repeated Sets of Back Squats. J Strength Cond Res. 2025 Jun 1;39(6):617-624. doi: 10.1519/JSC.0000000000005085. Epub 2025 Apr 23. PMID 40267419